CLINICAL TRIAL: NCT06679309
Title: Paving a Road Map for Integrated Care Evaluation in Canada: A Mixed Methods Evaluation for Patients With Complex Care Needs in Ontario and Alberta
Brief Title: ICP for Patients With Complex Care Needs in Ontario and Alberta, Canada
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: REB23-1442; 202211IS6 (Other: THINC Implementation Science Team Grants, CIHR)
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Health Care Quality, Access, and Evaluation
Keywords: integrated care; patient experience; provider experience; continuum of care; medical vulnerability; social determinants of health; psychosocial vulnerability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Integrated care pathway supported by the integrated care lead (Experimental): Enrolled patients in the ICP will then undergo more assessment by the Integrated Care Lead to develop a preliminary inventory of their needs for transitioning back to their health home. Patients will then be assigned an Integrated Care Lead with expertise in managing their particular needs. This will result in the development of a complex care plan that is co-designed with a patient's acute and community care team (eg: primary care, home care, community services, hospital medical team etc). This plan will be documented in Connect Care and incorporated into the discharge summary at the time of hospital discharge. (see Appendix 2)
  Calgary Zone Integrated Care Program will then provide:
  * Continuity of care with the assigned ICP team member(s) throughout their hospitalization and connection with community resources and services in the process of complex discharge planning.
  * Efficient use of healthcare resources by reducing duplication of services and systematically screening for unmet
  Interventions: Other: Integrated care plan

INTERVENTIONS:
Other: Integrated care plan — Complex care plan facilitated by the integrated care lead with 90 day follow-up, 24/7 phone support and connection with resources and services

SUMMARY:
The Integrated Care Pathway (ICP) model can reduce hospital readmissions and emergency department (ED) visits while improving continuity of care. This model was first developed at the University Health Network in Toronto, Ontario, and has been adapted for patients at high risk of readmission and with medical/social vulnerability admitted to general medical units in the hospitals in Calgary, Alberta. The study will evaluate the ongoing adaption and implementation of the ICP model in Calgary.

ICP patients will receive the following tenets of care:

1. Continuity of care - After determining the patient's inventory of needs, study participants will then be assigned to an ICP team member who will follow them throughout their hospitalization to support their discharge planning and to advocate for their needs in hospital.
2. Intensive Case Management - The ICL will liaise with hospital, primary care and community partners to develop a tailored complex care plan to support the patient's transition home. This will be documented in the hospital's electronic medical record (EMR) and incorporated into the discharge summary at the time of hospital discharge.
3. Post-discharge support

   * 24 hour access to phone support within the first 2 weeks of discharge from hospital, leveraging the ICP, community stakeholders and Healthlink from Alberta Health Services.
   * Long-term support and follow-up in the community up to 90 days with goal of implementing and adapting the complex care plan to help patients access services and manage their chronic health conditions.

The main study objectives are:

1. To adapt and implement the ICP in Calgary's 4 hospitals over a 3 year period.
2. To evaluate the implementation of the ICP in Calgary leveraging the Quintuple Aim Framework.

Methods:

Patients enrolled in ICP will be compared with comparator patients in control sites to evaluate the model's effectiveness.

Since the ICP is new to Calgary, the research team will be evaluating how well it performs compared to usual transitions in care by collecting data to learn about:

1. How patients and their caregivers experienced their time in hospital and transition home.
2. How healthcare providers feel about the ICP's impact on patient care.
3. The ICP's impact on patient health outcomes,
4. The use of hospital resources, and the cost of providing care.
5. The ICP's impact on equity, or fair access to healthcare resources and services.

DETAILED DESCRIPTION:
1.0 BACKGROUND Twenty percent of Canadian adults are living with multiple chronic diseases, and are among the highest users of the health system, with the poorest outcomes. Hospital admissions account for approximately 30% of all healthcare spending and are associated with a higher risk of death and complications. For example, older adults (over age 65) have a 6-fold increased risk of discharge to long-term care, and a 34.3-fold increased chance of dying in hospital. Furthermore, approximately 8.5% of acute care patients have a readmission within 30 days of their initial hospitalization. This is estimated to cost $1.8 billion and account for 11% of all acute care hospital costs. As such, there is an urgent need to develop models of care that address the root causes of the current reliance on hospitals, which is both an inefficient use of resources, and is associated with deleterious outcomes for the most vulnerable patients.

Prior to 2019, the Ontario Ministry of Health and Long-Term Care funded a consortium of pilot projects in Ontario to test integration of care initiatives that improve healthcare system sustainability and patient outcomes. Institutions using this model showed reduced mean length of stay by 1.26 days, emergency department (ED) visits or death at 30 days post discharge by 6%, readmission and death rates within 30 days post-discharge by 6%, mean total costs by $3035 within 90 days of admission.

Subsequently, the University Health Network (UHN) adapted the successful pathway from this initiative to create the Integrated Care Pathway (ICP) (see Appendix 1 in study protocol) in Toronto with the following services for individuals enrolled in the pathway:

1. Access to one care team- including connection to an Integrated Care lead during admission to hospital to create a complex transitional care plan that links with community services and primary care.
2. Access to one point of contact for support via a 24/7 phone line.
3. One shared electronic health record across acute care and home and community care.
4. Benefit from a flexible approach to funding that allows care to be personalized- this includes remote care monitoring and virtual care (where applicable).
5. Coordination of primary care, home and community-care and is supported by one funding source which follows the patient following discharge from hospital for up to 90 days (depending on patient need).

As of Fall 2022, 2220 patients were enrolled in UHN's ICP in multiple departments spanning several complex conditions. A mixed methods evaluation of the ICP among thoracic surgery patients demonstrated feasibility, minimal change in workload for front-line health care staff, qualitative improvements in patient experience, along with a 28% decreased length of stay, 45% reduction in ED visits and 33% reduction in hospital readmissions at 3 months following entry into the program. The program was spread to vascular and cardiovascular surgery, and in January 2022, to complex medical inpatients starting with congestive heart failure (CHF), chronic obstruction pulmonary disease (COPD) and COVID-19.

The proposed intervention is an adaptation of UHN's established Integrated Care Pathway (ICP) model of care for the Calgary Zone (see figure in Appendix 2). In Calgary, many of the essential components of the intervention are already established but operate in siloes. Over the past year, the Calgary ICP team has engaged multiple stakeholders across the continuum of care to develop a locally sustainable pathway that adheres to the principles of UHN's ICP, but leverages Calgary's strengths and fills existing care gaps.

2.0 OBJECTIVE: To evaluate the ongoing adaption and implementation of the ICP model in Calgary Zone

METHODS:

Target population: Patients admitted to a Calgary Hospital with:

1. medical vulnerability - includes multimorbidity (2+ medical conditions requiring ongoing monitoring, frailty, polypharmacy, high risk of readmissions/death)
2. psychosocial vulnerability - includes social, financial or behavioral challenges that impede a patient from accessing healthcare or other services without extra support

SUBJECT ENROLLMENT 4.1 Patient recruitment The nursing and/or research teams will systematically screen newly admitted patients to intervention sites' hospital medicine units (General Internal Medicine and Hospitalist Medicine) for inclusion / exclusion criteria (see above). This will require a waiver of consent for the initial screening to enable the team to screen all patients in order to identify potential candidates.

Patients deemed to be potentially eligible for the program will then be approached by the ICP team (either nurse or research assistant) to explain ICP and the research study, either verbally or with a short video. Patients expressing interest in the study will be asked to provide virtual and/or written informed consent using e-consent through REDCap (Research Electronic Data Capture, Vanderbilt University, Nashville, TN) and will be enrolled in the study.

4.2 Caregiver recruitment The ICL will identify caregivers of patients that consent to participate in the study, and provide them with information about the program/answer initial questions. If the caregiver expresses interest and meets inclusion criteria the research assistant/coordinator will assist in the informed consent process by reviewing the consent form with the caregiver, and obtaining written informed consent or electronic informed consent through REDCap.

4.3 Healthcare Provider (HCP) recruitment Members of the ICP clinical team and clinicians working alongside the ICP team at each study site will be identified and offered participation in the study by the research team. Similarly, patients' family doctors will be offered participation in the study. If the clinician agrees, the research assistant/coordinator will discuss the purpose of the study with them (including what data the investigators will be collecting from rural home hospital clinicians and why) and invite them to participate in surveys and semi-structured interviews. If the clinician agrees to enroll, the research assistant/coordinator will assist in the informed consent process by reviewing the consent form with the clinician to obtain written informed consent or electronic informed consent through REDCap.

PROCEDURES 5.1 Intervention Enrolled patients in the ICP will then undergo more assessment by the Integrated Care Lead to develop a preliminary inventory of their needs for transitioning back to their health home. Patients will then be assigned an Integrated Care Lead with expertise in managing their particular needs. This will result in the development of a complex care plan that is co-designed with a patient's acute and community care team (eg: primary care, home care, community services, hospital medical team etc). This plan will be documented in Connect Care and incorporated into the discharge summary at the time of hospital discharge. (see Appendix 2)

Calgary Zone Integrated Care Program will then provide:

* Continuity of care with the assigned ICP team member(s) throughout their hospitalization and connection with community resources and services in the process of complex discharge planning.
* Efficient use of healthcare resources by reducing duplication of services and systematically screening for unmet needs in order to systematically connect patients with the services and resources participants need when participants leave the hospital.
* 24 hour access to phone support within the first 2 weeks of discharge from hospital, leveraging the ICP, community stakeholders and Healthlink from Alberta Health Services
* Long-term support and follow-up in the community up to 90 days with goal of implementing and adapting the complex care plan to help patients access services and manage their chronic health conditions.

5.2 Evaluation Methods Procedures/ interventions The Integrated Care Pathway will not alter existing usual care standards, but will leverage and enhance existing processes for discharge planning and transitions of care. The ICP will be implemented over the course of 3 years at the four Calgary hospitals: the Foothills Medical Centre (FMC), Peter Lougheed Centre (PLC), South Health Campus (SHC), and the Rockyview General Hospital (RGH).

Enrolled patients in the ICP will then undergo more assessment by the Integrated Care Lead to develop a preliminary inventory of their needs for transitioning back to their health home. Patients will then be assigned an Integrated Care Lead with expertise in managing their particular needs. This will result in the development of a complex care plan that is co-designed with a patient's acute and community care team (eg: primary care, home care, community services, hospital medical team etc). This plan will be documented in Connect Care and incorporated into the discharge summary at the time of hospital discharge. (see Appendix 2)

Calgary Zone Integrated Care Program will then provide:

* Continuity of care with the assigned ICP team member(s) throughout their hospitalization and connection with community resources and services in the process of complex discharge planning.
* Efficient use of healthcare resources by reducing duplication of services and systematically screening for unmet needs in order to systematically connect patients with the services and resources participants need when participants leave the hospital.
* 24 hour access to phone support within the first 2 weeks of discharge from hospital, leveraging the ICP, community stakeholders and Healthlink from Alberta Health Services
* Long-term support and follow-up in the community up to 90 days with goal of implementing and adapting the complex care plan to help patients access services and manage their chronic health conditions.

5.2 Evaluation Methods This is a prospective multi-centre quasi-experimental study since the ICP will be rolled out at successive sites in Calgary over the next 2 years. Patient-level data will help evaluate the clinical intervention's impact on patient and caregiver outcomes and experience. Site-level data will be used to evaluate impact on the healthcare system. Sites will all serve as historical controls until the ICP is implemented at each site. At that point participants will then begin to contribute data as an intervention site in a stepped wedge non-randomized design.

5.2.1 Implementation and process evaluation

The investigators will perform a mixed methods evaluation using the QIF, which identiﬁes the following four phases with speciﬁc actions to guide implementation and evaluation to achieve quality improvement:

1. Establishment of a structure for ICP: Activities will be mapped out to identify key qualified individuals to take responsibility for implementation and help identify the structures and process of the ICP. The structures will be described as: 1) organizational supports, 2) team and clinical resources, 3) acute care partners, 4) primary care partners, 5) community partners and 6) IT infrastructure/minimum data set.
2. Implementation of ICP processes with the following assessment: a) uptake of ICP components (referral volume and acceptance to pathway, patient experience, secondary outcomes including timeliness of follow-up and community services) and provider experience with care provision.
3. Ongoing structure modifications once implementation begins: Activities include provision of technical supports, monitoring implementation and creating feedback mechanisms for progression. Provider adherence to ICP will be monitored to ensure relevance to end-user's needs. Baseline values will be determined in the first months using the Interrupted Time Series design. Acceptability of ICP will be measured for both processes and structures at patient, caregiver and provider levels. Qualitative data will provide contextual information related to implementation and will explore 1) participants' views and acceptability of ICP; and 2) aspects related to implementation, feasibility and usefulness of the program. Organizational structures such as 1) consistency of minimum data set and IT infrastructure; and 2) integration of ICP pathway use amongst providers will be assessed through documentation of organizational processes and a fidelity checklist.
4. Improving Future Applications: Activities will focus on learnings from experience (i.e., identification of facilitators and barriers for future scale and spread) and maintaining learnings across time. ICP maintenance goals include: 1) refining the set of core competencies and training program that instills these competencies; 2) establishing best practices for providers across care settings; 3) use of common infrastructures for record keeping and documentation of activities; 4) successful integration of ICP and community programs. In this final phase the investigators will document how aspects of the intervention are sustained or change over time and beyond their support period. This will be the foundational information for the toolkit that incorporates important program refinements identified in our evaluation. Once the structural components of the ICP have been established, the research team will work collaboratively to develop key education and training modules, which will be tailored to end-user groups (those with multimorbidity and older adults with complex care needs) in both acute and community care. These knowledge dissemination products (i.e., the toolkit) will be highly valuable in supporting the future spread of the program to additional sites and other chronic conditions beyond those currently identified.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS:

  1. Over 18 years of age
  2. Able to provide informed consent, or has substitute-decision-maker and is able to provide assent.
  3. Resides in Calgary Zone
  4. High risk of readmission and/or social vulnerability:

     * medical vulnerablility - includes multimorbidity (2+ medical conditions requiring ongoing monitoring, frailty, polypharmacy, high risk of readmissions/death)
     * psychosocial vulnerability - includes social, financial or behavioural challenges that impede a patient from accessing healthcare or other services without extra support
  5. Attached to primary care or has potential for access to health resources can be reasonably obtained in the short-term via access clinics or community agency follow-up.
  6. Community-dwelling

CAREGIVER

1. Informal caregiver (friend/family) of a patient enrolled in ICP (eg: provides support in form of care at home, transportation / going to appointments, managing finances etc)
2. Provides informed consent to participate in the study.

PROVIDERS

1. Healthcare professional working in the program, or having had a patient enrolled in the program within the past 3 months (eg: nurse, doctor, allied health professional etc)
2. Provides informed consent to participate in the study

Exclusion Criteria:

* 1) Patient characteristics:

  * Competent patient and/or substitute decision-maker who declines to provide informed consent to participate in ICP program
  * On Mental Health Form 1 / active psychosis / suicide risk / intoxication
  * Patients without valid health coverage data
  * Patients that are critically ill and likely to die in hospital

    2) Alternative care arrangements / pathways or not in catchment
  * Individuals being discharged to Supportive Living / Long-term care / rehabilitation
  * Patients requiring end-of-life care
  * Resides outside of Calgary Zone
  * In police custody

    3) Non-hospital medicine populations
  * Pediatric (17 years or younger)
  * Admitted to surgery, obstetrics/gynecology
  * Admitted to a psychiatric ward

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient experience | From enrollment to 90 days post-discharge
  Proportion of patients reporting a positive experience up to three months following discharge from an acute care hospital, as defined by having the following top box (positive) responses to seven patient experience questions from the Canadian Institute for Health Information (CIHI) Canadian Patient Experience Survey on Inpatient Care (CPES-IC) , a standardized and validated survey sent out by all hospitals in English and/or French (see Appendix for all questions). Response options include ordinal frequencies or binary responses to questions focused on communication and care coordination (e.g., "During this hospital stay, did doctors, nurses, or other hospital staff talk with you about whether you would have the help needed when you left hospital?"). The choice of top-box response to patient experience survey questions is being used to align with Canadian benchmarking and for comparison with HCAHPS patient experience survey questions for international representation ,.

SECONDARY OUTCOMES:
Re-admission | up to 3 months after discharge
  The proportion of patients which had a primary care or subspecialty visit, in the 7 days, 1 and 3 months after discharge will be estimated with the cumulative incidence, taking into account competing risks due to death and hospital readmission during this time.

OTHER OUTCOMES:
Quintuple Aim - a conceptual framework for evaluating quality of healthcare services developed by the Institute of Healthcare Improvement for evaluating new health programs | minimum 6 months post-implementation of ICP at all sites
  Quintuple Aim - a conceptual framework for evaluating quality of healthcare services developed by the Institute of Healthcare Improvement for evaluating new health programs.1 This framework has 5 domains for assessing quality of care: 1) patient experience (survey); 2) provider experience (survey and interview; 3) patient/population health outcomes (health-related quality of life at enrollment, discharge, 30 days), mortality during admission, 30 days, 90 days, 4) healthcare costs and utilization (% of patients with follow-up visits to primary care within 7, 14, 30 days; % of patients with outpatient visits with subspecialty care with 7 days and 1 month following discharge from hospital, measured seperately; Time to first home-care service following discharge; percentage with return to ED, or non-elective readmission to hospital, measured separately within 7 days and 1 month following discharege;overall cost of care) 5) equity (social determinants of health)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Grinman, MD FRCPC MPH, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Wandersman A, Duffy J, Flaspohler P, Noonan R, Lubell K, Stillman L, Blachman M, Dunville R, Saul J. Bridging the gap between prevention research and practice: the interactive systems framework for dissemination and implementation. Am J Community Psychol. 2008 Jun;41(3-4):171-81. doi: 10.1007/s10464-008-9174-z. PMID 18302018
- [Background] Nundy S, Cooper LA, Mate KS. The Quintuple Aim for Health Care Improvement: A New Imperative to Advance Health Equity. JAMA. 2022 Feb 8;327(6):521-522. doi: 10.1001/jama.2021.25181. No abstract available. PMID 35061006
- [Background] Meyers DC, Durlak JA, Wandersman A. The quality implementation framework: a synthesis of critical steps in the implementation process. Am J Community Psychol. 2012 Dec;50(3-4):462-80. doi: 10.1007/s10464-012-9522-x. PMID 22644083
- [Background] Steele Gray C, Zonneveld N, Breton M, Wankah P, Shaw J, Anderson GM, Wodchis WP. Comparing International Models of Integrated Care: How Can We Learn Across Borders? Int J Integr Care. 2020 Apr 1;20(1):14. doi: 10.5334/ijic.5413. PMID 32292312
- [Background] Kiran T, Wells D, Okrainec K, Kennedy C, Devotta K, Mabaya G, Phillips L, Lang A, O'Campo P. Patient and caregiver experience in the transition from hospital to home - brainstorming results from group concept mapping: a patient-oriented study. CMAJ Open. 2020 Mar 2;8(1):E121-E133. doi: 10.9778/cmajo.20190009. Print 2020 Jan-Mar. PMID 32127383
- [Background] Hunting G, Shahid N, Sahakyan Y, Fan I, Moneypenny CR, Stanimirovic A, North T, Petrosyan Y, Krahn MD, Rac VE. A multi-level qualitative analysis of Telehomecare in Ontario: challenges and opportunities. BMC Health Serv Res. 2015 Dec 9;15:544. doi: 10.1186/s12913-015-1196-2. PMID 26645639
- [Background] Hahn-Goldberg S, Huynh T, Chaput A, Krahn M, Rac V, Tomlinson G, Matelski J, Abrams H, Bell C, Madho C, Ferguson C, Turcotte A, Free C, Hogan S, Nicholas B, Oldershaw B, Okrainec K. Implementation, spread and impact of the Patient Oriented Discharge Summary (PODS) across Ontario hospitals: a mixed methods evaluation. BMC Health Serv Res. 2021 Apr 17;21(1):361. doi: 10.1186/s12913-021-06374-8. PMID 33865385
- [Background] Isaac T, Zaslavsky AM, Cleary PD, Landon BE. The relationship between patients' perception of care and measures of hospital quality and safety. Health Serv Res. 2010 Aug;45(4):1024-40. doi: 10.1111/j.1475-6773.2010.01122.x. Epub 2010 May 28. PMID 20528990
- [Background] Griffiths S, Stephen G, Kiran T, Okrainec K. "She knows me best": a qualitative study of patient and caregiver views on the role of the primary care physician follow-up post-hospital discharge in individuals admitted with chronic obstructive pulmonary disease or congestive heart failure. BMC Fam Pract. 2021 Sep 7;22(1):176. doi: 10.1186/s12875-021-01524-7. PMID 34488652
- [Background] Okrainec K, Chaput A, Rac VE, Tomlinson G, Matelski J, Robson M, Troup A, Krahn M, Hahn-Goldberg S. Raising the bar for patient experience during care transitions in Canada: A repeated cross-sectional survey evaluating a patient-oriented discharge summary at Ontario hospitals. PLoS One. 2022 Oct 4;17(10):e0268418. doi: 10.1371/journal.pone.0268418. eCollection 2022. PMID 36194600
- [Background] Okrainec K, Hahn-Goldberg S, Abrams H, Bell CM, Soong C, Hart M, Shea B, Schmidt S, Troup A, Jeffs L. Patients' and caregivers' perspectives on factors that influence understanding of and adherence to hospital discharge instructions: a qualitative study. CMAJ Open. 2019 Jul 18;7(3):E478-E483. doi: 10.9778/cmajo.20180208. Print 2019 Jul-Sep. PMID 31320331